CLINICAL TRIAL: NCT03075241
Title: Z-Drugs for the Treatment of Sleep Disorders in Alzheimer's Disease: a Randomized, Triple-blind, Placebo-controlled Study
Brief Title: Z-Drugs for Sleep Disorders in Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Einstein Francisco de Camargos, Principal Investigator, Brasilia University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZOLP-001
Record Dates: First submitted 2017-03-05; First posted 2017-03-09 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Sleep; Sleep Disorders; Insomnia; Alzheimer's Disease
Keywords: Sleep Disturbances; Alzheimer Disease; Insomnia; Z-Drugs; Treatment
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders; Alzheimer Disease; Parasomnias | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Zolpidem (Experimental): Study group will receive zolpidem 10mg capsules, 10pm (before bedtime) for 14 nights
  Interventions: Drug: Zolpidem
- Zoplicone (Experimental): Study group will receive zoplicone 7.5mg capsules, 10pm (before bedtime) for 14 nights
  Interventions: Drug: Zoplicone
- Placebo (Placebo Comparator): Study group will receive inactive or inert capsules, which will be used as a comparator, 10pm (before bedtime) for 14 nights
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zolpidem — Zolpidem tablets, 10mg, 10pm (before bedtime) for 14 nights
  Arms: Zolpidem
Drug: Zoplicone — Zoplicone tablets, 7.5mg, 10pm (before bedtime) for 14 nights
  Arms: Zoplicone
Drug: Placebo — Inactive or inert pill which will be used as a comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Zolpidem and Zoplicone are efective in the treatment of sleep disorders in Alzheimer's disease (AD)

DETAILED DESCRIPTION:
Sleep disorders (SD) affects 35 to 50 percent of patients with AD. These disorders often make caring for patients at home very difficult. Zolpidem and Zoplicone are prescribed drugs for sleep disorder in AD patients.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* Diagnosis of probable Alzheimer's disease (AD) by National Institute of Neurological and Communicative Disorders and Stroke / the Alzheimer's Disease and Related Disorders Association Criteria
* Hachinski Ischemia Scale less than 5
* Mini-Mental State Examination score of 0 to 26
* Actigraph evidence of a mean time immobile of less than 7 hours per night based on at least 7 nights of complete actigraph data collected over a single week
* Four-week history of sleep disorder behaviors, occurring at least once weekly, as reported by the caregiver using the Neuropsychiatric Inventory (NPI) Nighttime Behavior scale
* Sleep disturbance observed was not present before the diagnosis of AD
* Other co-morbidities, especially delirium, depression, chronic pain and medication use may be present, but do not cooperate in the primary symptoms
* Computed tomography or magnetic resonance imaging since the onset of memory problems showing no more than 1 lacunar infract in a nonstrategic area and no clinical events suggestive of stroke or other intracranial disease or normal
* Stable medications for 4 weeks prior to the screening visit
* Having a mobile upper extremity to which to attach an actigraph
* Residing with a responsible spouse, family member, or professional caregiver who is present during the night and would agree to assume the role of the principle caregiver for the 3-week protocol
* Ability to ingest oral medication and participate in all scheduled evaluations

Exclusion Criteria:

* Sleep disturbance associated with an acute illness, delirium or psychiatric disease
* Clinically significant movement disorder, such as akinesia, that would affect actigraphic differentiation of sleep and wakefulness
* Severe agitation
* Unstable medical condition
* Discontinuation of psychotropic or sleep medication within 2 weeks of the screening visit
* Patient unwilling to maintain caffeine abstinence after 2:00pm for the duration of the protocol
* Patient unwilling to comply with the maximum limit of 2 alcoholic drinks per day, and only 1 alcoholic drink after 6:00pm for the duration of the protocolo
* Prior use of zolpidem/zoplicone for the treatment os sleep disturbances
* Caregiver deemed to be unreliable to supervise the wearing of the actigraph, to administer study capsules at the proper time, to maintain the sleep diary, or to bring the patient to the scheduled visits

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Nighttime Total Sleep Time | Baseline, 14 days follow-up
  Mean Total Sleep Time (in minutes) during the 12h nocturnal period (8:00pm-8:00am) after 2 weeks under treatment

SECONDARY OUTCOMES:
Daytime Total Sleep Time | Baseline, 14 days follow-up
  Daytime Total Sleep Time (in minutes) during the 12h daytime period (8:00am-8:00pm) after 2 weeks under treatment
Ratio of daytime to nighttime sleep | Baseline, 14 days follow-up
  Daytime Total Sleep Time / Nighttime Total Sleep Time
Nighttime Wake after Sleep Onset | Baseline, 14 days follow-up
  Nighttime Wake after Sleep Onset (in minutes) during the 12h nocturnal period (8:00pm-8:00am) after 2 weeks under treatment
Proportion of sleep time at nighttime | Baseline, 14 days follow-up
  Proportion of sleep time (%) during the 12h nocturnal period (8:00pm-8:00am) after 2 weeks under treatment
Proportion of patients with gain of at least 30 minutes in Total Sleep Time | Baseline, 14 days follow-up
  Proportion of patients with gain of at least 30 minutes in Total Sleep Time after 2 weeks under treatment
Differences between sleep efficiency between the two treatments. | Baseline, 14 days follow-up
  Analyze possible differences between sleep efficiency between the two treatments after 2 weeks under treatment
Nighttime Number of Awakenings | Baseline, 14 days follow-up
  Change in scores of nighttime number of awakenings from baseline to intervention weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luciana L. Louzada, MD, MsC, Principal Investigator — Brasilia University - Brasilia's University Hospital - Geriatric Medical Center
Locations (1):
- Geriatric Medical Centre, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Louzada LL, Machado FV, Quintas JL, Ribeiro GA, Silva MV, Mendonca-Silva DL, Goncalves BSB, Nobrega OT, Camargos EF. The efficacy and safety of zolpidem and zopiclone to treat insomnia in Alzheimer's disease: a randomized, triple-blind, placebo-controlled trial. Neuropsychopharmacology. 2022 Jan;47(2):570-579. doi: 10.1038/s41386-021-01191-3. Epub 2021 Oct 11. PMID 34635802